CLINICAL TRIAL: NCT07056426
Title: Comparison of the Effectiveness of Extracorporeal Shock Wave Therapy and Deep Tissue Massage in Individuals With Medial Tibial Stress Syndrome
Brief Title: Comparison of ESWT and Deep Tissue Massage in Individuals With Medial Tibial Stress Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Murat Akıncı, Pricipal Investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTSS01
Record Dates: First submitted 2025-06-11; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Medial Tibial Stress Syndrome
Keywords: Medial Tibial Stress Syndrome; Shin Splint; ESWT; Deep Tissue Massage
MeSH Terms: conditions — Medial Tibial Stress Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Experimental): ESWT will be applied once weekly for four sessions, delivering 2000 pulses per session at 2.5 bar pressure and 8 Hz frequency using radial shock waves. Each session's energy flux density is about 200 mJ/mm². The patient will lie supine, with ultrasound gel applied to the medial tibial area. Shock waves will be delivered in a circular motion from medial to lateral, focusing on the most sensitive and painful spot, covering an area approximately 2-4 cm wide and 4-8 cm long.
  Interventions: Other: Exercises; Other: ESWT
- Deep Tissue (Experimental): The deep tissue massage will be performed with the patient lying on their side, affected leg on top and knee flexed at about 45 degrees, with the medial tibia facing upward. After applying petroleum jelly, palpation will locate the sensitive medial tibial line. The massage begins with 4-5 superficial strokes along this line, followed by 2-3 deeper strokes to assess muscle tone and sensitivity. Moderate pressure is then applied with the thumb perpendicular to the tibial line, starting just above the medial malleolus and moving slowly toward the medial tibial plateau, before shifting one finger width posteriorly to massage upward along the soleus muscle. These steps are repeated 6-8 times, each lasting 10-15 seconds, with pressure adjusted to a pain level of 7-8 on the Visual Analog Scale (VAS). A 10-second rest is given between applications, and the session ends with 4-5 superficial strokes.
  Interventions: Other: Exercises; Other: Deep Tissue Massage

INTERVENTIONS:
Other: Exercises — Joint mobilization exercises:
  -Active ankle range of motion exercises
  Ankle strengthening with resistance band (Thera-band®):
  * Resisted dorsiflexion
  * Resisted plantar flexion
  * Resisted inversion
  * Resisted eversion
  * Leg muscle strengthening exercises:
  * Heel raises (standing)
  * Heel raises (sitting)
  * Toe raises (standing)
  * Toe raises (sitting)
  Hip and pelvis stabilizer muscle strengthening exercises:
  * Pelvic bridge
  * Side leg lifts with hip and knee at 0°
  * Side leg lifts with hip and knee at 90°
  Stretching exercises:
  * Calf stretch with towel
  * Gastrocnemius stretch (standing)
  * Soleus stretch (standing)
  * Anterior compartment leg stretch
  These exercises will be applied three times a week in 40-minute sessions, for a total of 12 sessions.
Other: ESWT — The Extracorporeal Shock Wave Therapy (ESWT) will be administered once a week for a total of four sessions. Each session will deliver 2000 pulses at a pressure of 2.5 bar and a frequency of 8 Hz using radial shock wave technology. The total energy flux density per session is planned to be approximately 200 mJ/mm².
  Patients will be positioned in a supine lying position during the treatment. A generous amount of ultrasound gel will be applied to the medial tibial border and surrounding tissues to ensure effective transmission of shock waves and patient comfort.
  The application of shock waves will follow the clinical focusing principle: treatment will start from the point of greatest tenderness and maximal pain on the medial tibial border, progressing in a circular motion from medial to lateral. The treatment area will typically cover a region approximately 2-4 cm in width and 4-8 cm in length.
  Arms: ESWT
Other: Deep Tissue Massage — The deep tissue massage begins with the patient lying on their side, the affected leg on top, knee flexed at about 45 degrees, and the medial surface of the tibia facing upward. The sensitive line along the medial tibia is identified by palpation, and the area is prepared with petroleum jelly. The massage starts with 4-5 superficial strokes along the medial calf using the palm, followed by 2-3 deep strokes to assess muscle tone and patient tolerance. Moderate pressure is applied with the thumb perpendicular to the tibial line, moving slowly from just above the medial malleolus toward the medial tibial plateau. Then, the thumb shifts one finger width posteriorly and moves upward along the soleus muscle with similar pressure. These two steps are repeated 6-8 times, each lasting 10-15 seconds, with pain adjusted to 7-8 on the VAS scale. A 10-second rest is given between applications, and the massage ends with 4-5 superficial strokes.
  Arms: Deep Tissue

SUMMARY:
This study, titled "Comparison of the Effectiveness of Extracorporeal Shock Wave Therapy and Deep Tissue Massage in Individuals with Medial Tibial Stress Syndrome (MTSS)," is designed as a prospective, randomized controlled trial with two parallel groups. The research will be conducted at the Sports Health Laboratory of the Ankara Bilkent City Hospital, Department of Physical Medicine and Rehabilitation.

The study population will consist of individuals who meet the diagnostic criteria for MTSS and present to the Sports Medicine outpatient clinic.

All participants will undergo an exercise program recommended in the literature for the treatment of MTSS. Participants will be randomly assigned into two groups using a sealed-envelope method. One group will receive deep tissue massage in addition to the exercise program, while the other group will receive extracorporeal shock wave therapy (ESWT) alongside the exercises. Additionally, all participants will be treated with conventional transcutaneous electrical nerve stimulation (TENS) at 100 Hz for pain control.

Initial assessments, randomization, treatment applications (TENS, exercise, deep tissue massage, and ESWT), and outcome evaluations will be performed by different members of the research team. Outcome assessments will be conducted in a blinded manner to ensure objectivity regarding treatment allocation.

DETAILED DESCRIPTION:
Medial Tibial Stress Syndrome (MTSS) is often inadequately treated with standard methods. This study aimed to investigate the effects of deep tissue massage, considered as an alternative and adjunct treatment method, on pain and functional capacity in individuals diagnosed with MTSS, and to compare its efficacy with Extracorporeal Shock Wave Therapy (ESWT), a widely accepted treatment. The study was designed as a prospective, parallel-group trial and conducted at a sports health laboratory affiliated with a physical therapy and rehabilitation hospital. The study population consisted of patients who met MTSS diagnostic criteria and presented to a sports medicine outpatient clinic.

MTSS is characterized by pain along the medial border of the tibia during running or walking, with a gradual onset unrelated to traumatic events, and diffuse pain upon palpation along the medial tibial border. It is one of the most common overuse injuries affecting a significant portion of the athletic population. Although the exact pathophysiology of MTSS is not fully understood, pain is thought to originate from inflammation at the periosteal-fascial junction or enthesis area, involving only soft tissues without bone stress reactions or fractures; however, bone involvement may coexist and exacerbate pain.

Various treatment approaches have been proposed for MTSS, including rest, activity modification, exercise programs, ESWT, and injections. Limited studies exist evaluating the efficacy of radial ESWT, which have shown improved recovery and return-to-sport rates compared to control groups. Nevertheless, ESWT has been insufficient for some patients, highlighting the need for alternative treatments. While the soleus muscle is generally considered the primary contributor to MTSS, the flexor digitorum longus and deep leg fascia also play roles due to their origins on the medial tibia. Deep tissue massage has been effective in plantar heel pain but lacks sufficient evidence in MTSS patients.

The purpose of this study was to assess the effect of deep tissue massage (targeting the soleus, flexor digitorum longus, and deep leg fascia) on pain in individuals with MTSS and to compare it with ESWT. A pilot study was planned with a total of 22 participants (11 per group), based on an estimated large effect size (Cohen's d=1.30). Participants received either ESWT or deep tissue massage in addition to transcutaneous electrical nerve stimulation (TENS) and a standard exercise program. The exercise program consisted of 12 sessions of 40 minutes each, three times per week. Both ESWT and deep tissue massage were applied once weekly for four sessions. ESWT parameters included 2000 pulses per session, 2.5 bar pressure, 8 Hz frequency, and an energy flux density of approximately 200 mJ/mm². Deep tissue massage was performed with the patient lying on their side, knee flexed at 45 degrees, applying moderate pressure along the medial tibial line. Pain during massage was maintained at 7-8 on the Visual Analog Scale (VAS), with repeated 10-15 second applications.

The study duration was planned for one year following ethical approval, with recruitment starting in February 2025 and completion aimed for December 2025. Inclusion criteria were age over 18, recreational or professional athletes, diagnosed with MTSS as defined, and symptoms persisting for at least 3 weeks without any exclusion criteria. Exclusion criteria included presence of stress fractures or other fractures, history of chronic exertional compartment syndrome, previous ESWT or deep tissue massage for MTSS, rheumatologic diseases, local infection or tumor in the treatment area, pregnancy, bleeding disorders, advanced osteoarthritis of the ipsilateral knee or ankle, recent local injections, or prior knee/ankle surgery. Participants had the right to withdraw from the study at any time.

Outcome measures included demographic data collection before treatment and assessments at baseline, immediately after treatment, and at 8 weeks. Pain intensity was measured using the VAS during rest and exercise over the previous week. The painful area along the tibial border was measured in length. The Foot and Ankle Ability Measure (FAAM) assessed changes in physical function via self-reported questionnaires. Participants completed a treadmill test at a fixed speed of 10 km/h for 2000 meters, recording pain onset distance and pain levels at test completion or termination. The navicular drop test evaluated the medial longitudinal arch height difference between sitting and standing positions. The Foot Posture Index assessed foot posture across multiple segments using six criteria rated on a Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age,
* Those who participate in recreational or professional level sports,
* Those diagnosed with MTSS

Exclusion Criteria:

* Those with fracture findings, including radiological stress fractures,
* Those with a history of chronic exercise-related compartment syndrome,
* Those who have previously received ESWT (extracorporeal shock wave therapy) or deep tissue massage treatment for MTSS,
* Those with rheumatologic diseases (such as rheumatoid arthritis, widespread polyarthritis, etc.),
* Those with local infection or tumor in the treatment area,
* Pregnant women,
* Those with bleeding disorders,
* Those with advanced-stage ipsilateral knee and ankle osteoarthritis (defined by severe joint space narrowing, joint sclerosis, and periarticular osteophytes),
* Those who have received local injection (e.g., corticosteroids) in the treatment area within the last 3 months,
* Those who have previously undergone knee or ankle surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Day 0 (pre-treatment) and Week 3 (post-treatment)
  The intensity of pain in the medial region of the tibia will be measured by the Visual Analog Scale.
FAAM | Day 0 (pre-treatment) and Week 3 (post-treatment)
  Foot and Ankle Ability Measure: It is a self-reported scale developed to assess changes in physical function in individuals with musculoskeletal disorders of the foot, ankle, and lower leg, consisting of 29 Likert-type questions scored from 0 to 4 across daily living (21 items) and sports (8 items) subscales, with higher scores indicating better function, and includes additional questions scoring current function from 0 to 100, where 100 represents pre-injury function and 0 indicates inability to perform any normal daily activities.
Pain Area | Day 0 (pre-treatment) and Week 3 (post-treatment)
  The length of the painful area along the tibia will be recorded in centimeters.

SECONDARY OUTCOMES:
Pain with Activity | Day 0 (pre-treatment) and Week 3 (post-treatment)
  Pain levels during running at 10 km/h on a treadmill will be recorded, with the test ending either when the patient chooses to stop due to pain or after 2000 meters, and changes in pain on a 1-10 scale will be documented (e.g., pain of 3/10 occurred at 153 meters).

OTHER OUTCOMES:
Navicular Drop Test | Day 0 (pre-treatment) and Week 3 (post-treatment)
  The medial longitudinal arch height will be assessed with this test. While the patient is seated without bearing weight on the foot, the height of the navicular tuberosity from the ground will be marked and recorded on a white card. Then, with the patient standing upright and bearing equal weight on both feet, the height of the navicular tuberosity from the ground will be measured again, and the difference between the two measurements will be calculated. A difference of less than 5 mm indicates a supinated foot, 5-9 mm indicates a neutral foot, and greater than 9 mm indicates a pronated foot.
Foot Posture Index | Day 0 (pre-treatment) and Week 3 (post-treatment)
  It allows for a multiplanar, multi-segment assessment of foot posture. Six items are scored on a five-point Likert scale from +2 to -2 and summed: palpation of the talar head, inclination below and above the lateral malleolus, position of the calcaneus in the frontal plane (varus/valgus), bulging in the talonavicular joint area, structure of the medial longitudinal arch, and forefoot abduction/adduction relative to the rearfoot.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)